CLINICAL TRIAL: NCT02117258
Title: Randomized Phase II Study of Gemcitabine Plus Z-360 in Metastatic Pancreatic Adenocarcinoma Compared With Gemcitabine Plus Placebo ( ZIPANG Study )
Brief Title: Z-360 Plus GEM in Subjects With Metastatic Pancreatic Adenocarcinoma
Acronym: ZIPANG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z-360-01
Record Dates: First submitted 2014-04-07; First posted 2014-04-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Z-360, Pancreatic cancer, Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Z-360

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Z-360 60mg+Gemcitabine (Experimental): Z-360 60 mg will be taken orally, twice daily (BID) after a meal.
  Interventions: Drug: Z-360
- Z-360 120mg+Gemcitabine (Experimental): Z-360 120 mg will be taken orally, twice daily (BID) after a meal.
  Interventions: Drug: Z-360
- Z-360 240mg+Gemcitabine (Experimental): Z-360 240 mg will be taken orally, twice daily (BID) after a meal.
  Interventions: Drug: Z-360
- Placebo+Gemcitabine (Placebo Comparator): Placebo will be taken orally, twice daily (BID) after a meal.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Z-360 — Gemcitabine (1,000 mg/m^2) will be given by 30-minute intravenous infusion on Day 1, 8, and 15 followed by a one week rest in all 28-day Cycles, while Z-360 (60, 120 or 240 mg) will be taken orally, twice daily (BID) after a meal. Dosing will continue until the patient fulfills the withdrawal criteria.
  Arms: Z-360 120mg+Gemcitabine; Z-360 240mg+Gemcitabine; Z-360 60mg+Gemcitabine
Drug: Placebo — Gemcitabine (1,000 mg/m^2) will be given by 30-minute intravenous infusion on Day 1, 8, and 15 followed by a one week rest in all 28-day Cycles, while placebo will be taken orally, twice daily (BID) after a meal. Dosing will continue until the patient fulfills the withdrawal criteria.
  Arms: Placebo+Gemcitabine

SUMMARY:
The primary objective of this study is to compare the efficacy of GEM plus Z-360 versus GEM plus placebo on the overall survival (OS) in subjects with metastatic Pancreatic Adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects with histological or cytological evidence of metastatic Pancreatic Adenocarcinoma, Measurable disease or non-measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version criteria
* 2. Subjects with a life expectancy of at least 12 weeks,
* 3. Subjects with an Eastern cooperative oncology group performance status (ECOG PS) of 0, 1 or 2,
* 4. Subjects with the following adequate organ functions:

  * White blood cell count ≥3,000/μL (or absolute neutrophil count ≥1,500/μL) and ≤ 12,000/μL ,
  * Platelet count ≥100.0 × 10^9/L,
  * Hemoglobin ≥9.0 g/dL,
  * Serum creatinine ≤1.5 × the upper limit normal (ULN),
  * Total bilirubin ≤2.0 × ULN,
  * Serum aspartate transaminase levels ≤3.0 × ULN (≤5.0 × ULN in presence of liver metastases), and
  * Serum alanine aminotransferase levels ≤3.0 × ULN (≤5.0 × ULN in presence of liver metastases).

Exclusion Criteria:

* Subjects received the following previous therapies for Pancreatic Adenocarcinoma:

  * Surgery within the 4 weeks prior to randomization,
  * Radiation and chemoradiation within the 12 weeks prior to randomization,
  * Radiation for pain relief within the 4 weeks prior to randomization,
  * Gemcitabine used as a neoadjuvant or an adjuvant on surgery within the 24 weeks prior to randomization,
  * Chemotherapy except GEM used as an adjuvant on surgery within the 4 weeks prior to randomization,
  * Gemcitabine ≥600 mg/m^2 as sensitizer for chemoradiation,
  * Gemcitabine <600 mg/m^2 as sensitizer for chemoradiation within the 12 weeks prior to randomization,
  * Gemcitabine used for systemic chemotherapy, or
  * Systemic chemotherapies except GEM within the 4 weeks prior to randomization.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Approximately 24 months

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 24 months
Time to Treatment Failure | Approximately 24 months
Quality of Life | Approximately 24 months
Safety parameters | Approximately 24 months
  Incidence of SAEs and AEs, laboratory test results, vital signs, ECG results and physical examination findings
Pharmacokinetics | Day1
  To characterize the plasma pK of Z-360 when given in combination with GEM
Response Rate | Approximately 24 months
Benefit Rate | Approximately 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- Zeria Investigative sites, Japan, Japan
- Zeria Investigative Sites, Korea, South Korea
- Zeria Investigative Sites, Dawan, Taiwan